CLINICAL TRIAL: NCT03912909
Title: Effects of SGLT-2 Inhibition on Sympathetic Nervous System Activity in Humans
Brief Title: Effects of Sodium-glucose Co-transporter-2( SGLT-2 ) Inhibition on Sympathetic Nervous System Activity in Humans
Acronym: EMPA-SNS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Perth Hospital (Other)
Responsible Party: Principal Investigator, Dr Markus Schlaich, Principal Investigator, Royal Perth Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: REG 16-157
Record Dates: First submitted 2018-10-23; First posted 2019-04-11 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome; Type 2 Diabetes Mellitus; Obesity
Keywords: Metabolic Syndrome; Central sympathetic nervous system; Sodium-glucose co-transporter-2 (SGLT2); Blood Pressure
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Obesity | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Active Comparator): Empagliflozin 10mg daily or placebo
  Interventions: Drug: Empagliflozin Oral Tablet [Jardiance]; Drug: Placebo Oral Tablet
- Phase2 (Placebo Comparator): Empagliflozin 10mg daily or placebo
  Interventions: Drug: Empagliflozin Oral Tablet [Jardiance]; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin Oral Tablet [Jardiance] — Participants will be randomly assigned to receive either Empagliflozin 10mg/daily or Placebo and will later receive the alternate treatment. As the study is double blind neither the participant nor the study personnel will be aware of which treatment is currently being tested to avoid any effect this may have on the results. The two 4-week treatment phases will be separated by a 4-week wash out (drug-free) period. The study will consist of a total of 5 visits conducted over approximately 18 weeks; one screening visit, one baseline visit, 1 short visit at the start of the second treatment phase and 2 comprehensive testing visits, each at the end of the two treatment phases
Drug: Placebo Oral Tablet — Participants will be randomly assigned to receive either Empagliflozin 10mg/daily or Placebo and will later receive the alternate treatment. As the study is double blind neither the participant nor the study personnel will be aware of which treatment is currently being tested to avoid any effect this may have on the results. The two 4-week treatment phases will be separated by a 4-week wash out (drug-free) period. The study will consist of a total of 5 visits conducted over approximately 18 weeks; one screening visit, one baseline visit, 1 short visit at the start of the second treatment phase and 2 comprehensive testing visits, each at the end of the two treatment phases

SUMMARY:
This study is designed to investigate whether the sodium-glucose co-transporter-2 (SGLT-2) inhibitor Empagliflozin reduces sympathetic nervous system (SNS) activity in humans.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo controlled, cross-over study. Participants will be randomly assigned to receive either Empagliflozin 10mg/daily or Placebo and will later receive the alternate treatment.

Comprehensive testing will occur after each 4 week treatment phase and will include assessment of muscle sympathetic nerve activity, cardiac and renal noradrenaline spillover to assess organ specific SNS activity.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 -65 years
* (Body Mass Index) BMI≥30kg/m2
* Currently weight stable (+/- 3% in previous 6-12 months and not on any specific exercise or dietary program)
* Metabolic syndrome (defined as having: obesity (BMI ≥30kg/m2 ) plus any two of the following four factors: Elevated triglycerides (Triglyceride≥ 1.7mmol/L), Reduced HDL (High - density lipoprotein) cholesterol (<1.0mmol/L in males, <1.3mmol/L in females), Elevated clinic systolic (Blood Pressure) BP ≥130 or diastolic BP ≥85mmHg, Fasting glucose ≥5.6mmol/L or type 2 diabetes.
* office BP for screening purposes ≤160/90mmHg
* drug naïve for at least 6 weeks prior to baseline assessment

Exclusion Criteria:

* Grade 2-3 hypertension (systolic office BP >160, diastolic office BP >100 mmHg)
* Secondary causes of hypertension
* CKD (Chronic kidney disease) stage 4-5 {(estimated glomerular filtration) eGFR<30ml/min}
* Heart failure NYHA (New York Heart Association) class II-IV
* Recent CV (cardiovascular) event (acute myocardial infarction, acute coronary syndrome, stroke or transient ischaemic attack within the previous six months)
* unstable psychiatric condition
* medication such as corticosteroids, several antidepressants and antipsychotics
* Female participants of childbearing potential must have a negative pregnancy test prior to treatment

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in cardiac sympathetic nerve activity | 18 weeks
  Cardiac sympathetic nerve activity assessed by cardiac noradrenaline spillover
Reduction in renal sympathetic nerve activity | 18 weeks
  Renal sympathetic nerve activity assessed by renal noradrenaline spillover
Reduction in muscle sympathetic nerve activity | 18 weeks
  Muscle sympathetic nerve activity assessed by microneurography

SECONDARY OUTCOMES:
Reduction in ambulatory BP (blood pressure) | 18 weeks
  Blood Pressure assessed by ambulatory blood pressure monitoring
Reduction in central Blood Pressure | 18 weeks
  central Blood Pressure assessed by Sphygmocor XCEL
Change in urinary sodium excretion | 18 weeks
  Urinary sodium excretion assessed in a 24 hour urine sample
Change in glycemic control | 18 weeks
  Glycemic control as assessed by an oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, MD,FAHA,FESC, Principal Investigator — Royal Perth Hospital
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared to maintain anonymity and confidentiality of the participants

REFERENCES:
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Hall JE, Jones DW, Kuo JJ, da Silva A, Tallam LS, Liu J. Impact of the obesity epidemic on hypertension and renal disease. Curr Hypertens Rep. 2003 Oct;5(5):386-92. doi: 10.1007/s11906-003-0084-z. PMID 12948431
- [Background] Esler M, Straznicky N, Eikelis N, Masuo K, Lambert G, Lambert E. Mechanisms of sympathetic activation in obesity-related hypertension. Hypertension. 2006 Nov;48(5):787-96. doi: 10.1161/01.HYP.0000242642.42177.49. Epub 2006 Sep 25. No abstract available. PMID 17000932
- [Background] Straznicky NE, Grima MT, Sari CI, Karapanagiotidis S, Wong C, Eikelis N, Richards KL, Lee G, Nestel PJ, Dixon JB, Lambert GW, Schlaich MP, Lambert EA. The relation of glucose metabolism to left ventricular mass and function and sympathetic nervous system activity in obese subjects with metabolic syndrome. J Clin Endocrinol Metab. 2013 Feb;98(2):E227-37. doi: 10.1210/jc.2012-3277. Epub 2012 Dec 27. PMID 23271752
- [Background] Straznicky NE, Lambert EA, Grima MT, Eikelis N, Richards K, Nestel PJ, Dawood T, Masuo K, Sari CI, Dixon JB, Esler MD, Paul E, Schlaich MP, Lambert GW. The effects of dietary weight loss on indices of norepinephrine turnover: modulatory influence of hyperinsulinemia. Obesity (Silver Spring). 2014 Mar;22(3):652-62. doi: 10.1002/oby.20614. Epub 2013 Dec 6. PMID 23997009
- [Background] Schlaich MP, Kaye DM, Lambert E, Sommerville M, Socratous F, Esler MD. Relation between cardiac sympathetic activity and hypertensive left ventricular hypertrophy. Circulation. 2003 Aug 5;108(5):560-5. doi: 10.1161/01.CIR.0000081775.72651.B6. Epub 2003 Jul 7. PMID 12847071
- [Background] Ziegler D, Weise F, Langen KJ, Piolot R, Boy C, Hubinger A, Muller-Gartner HW, Gries FA. Effect of glycaemic control on myocardial sympathetic innervation assessed by [123I]metaiodobenzylguanidine scintigraphy: a 4-year prospective study in IDDM patients. Diabetologia. 1998 Apr;41(4):443-51. doi: 10.1007/s001250050928. PMID 9562349
- [Background] Sverrisdottir YB, Jansson LM, Hagg U, Gan LM. Muscle sympathetic nerve activity is related to a surrogate marker of endothelial function in healthy individuals. PLoS One. 2010 Feb 17;5(2):e9257. doi: 10.1371/journal.pone.0009257. PMID 20174639
- [Background] Mahfoud F, Schlaich M, Kindermann I, Ukena C, Cremers B, Brandt MC, Hoppe UC, Vonend O, Rump LC, Sobotka PA, Krum H, Esler M, Bohm M. Effect of renal sympathetic denervation on glucose metabolism in patients with resistant hypertension: a pilot study. Circulation. 2011 May 10;123(18):1940-6. doi: 10.1161/CIRCULATIONAHA.110.991869. Epub 2011 Apr 25. PMID 21518978